CLINICAL TRIAL: NCT01647750
Title: Study of Optimal Replacement of Thyroxine in the Elderly (SORTED) SORTED 1 - a Randomised Controlled Trial (Pilot Study), SORTED 2 - Qualitative Interviews, SORTED 3 - Retrospective Cohort
Brief Title: Study of Optimal Replacement of Thyroxine in the Elderly
Acronym: SORTED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5863; PB-PG-0610-22139 (Other Grant/Funding Number: National Institute for Health Research Research for patient Benefit); 2011-004425-27 (EudraCT Number); ISRCTN16043724 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2012-07-16; First posted 2012-07-24 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lower dose of levothyroxine (Other): Participants may be randomised to receive a lower dose of levothyroxine (lower than their usual dose) to achieve a target TSH level of 4.1 - 8.0 mU/L
  Interventions: Drug: Levothyroxine
- Standard dose of levothyroxine (Other): Patients may be randomised to receive their usual dose of levothyroxine (target TSH level 0.4 - 4.0 mU/L)
  Interventions: Drug: Levothyroxine

INTERVENTIONS:
Drug: Levothyroxine — Participants in the lower dose arm of the study will receive a lower dose of levothyroxine than their usual dose
  Arms: Lower dose of levothyroxine
Drug: Levothyroxine — Participants in the standard dose of treatment will receive their usual dose of levothyroxine
  Arms: Standard dose of levothyroxine

SUMMARY:
All patients with hypothyroidism are currently treated the same way, regardless of age. The investigators want to look at whether people aged 80 years or older would benefit from being treated with lower doses of levothyroxine. There are three reasons why the investigators think this could be beneficial, but this is not yet proven:

1. Some older people with hypothyroidism may have few symptoms.
2. Doctors look at the amount of Thyroid Stimulating Hormone (TSH) in the patient's blood to decide the dose of Thyroxine received. The standard "normal" TSH range used to determine the dose of levothyroxine is from younger people. The investigators wonder whether this is appropriate to all age ranges particularly as the investigators know that older people may normally have higher TSH values.
3. If TSH levels are too low there may be a slight increased risk of problems such as brittle bones or an irregular heartbeat.

The best way to test whether older people benefit from lower doses of levothyroxine is by a large clinical trial. Before the investigators can do this, the investigators need to run a smaller clinical trial called a "pilot study" (SORTED 1) to examine whether this is practical and acceptable. The pilot study aims to recruit 50 patients with hypothyroidism aged 80 or above.

Participants will be randomly allocated to receive their routine or lower dose of levothyroxine. Follow-up will be conducted over approximately 25 weeks.

The investigators also propose a qualitative study (SORTED 2) to specifically understand patient's willingness to take part in a RCT and participant's experience of the intervention.

Finally, the investigators propose a retrospective cohort study of 400 treated hypothyroid patients aged 80 years or more registered in 2008 in Primary Care Practices with the aim of studying outcomes after 4 years. The cohort study will collect data required to inform a sample size calculation for a future full study where the primary outcome will be 4 year mortality.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females aged 80 years or older
* Diagnosed with hypothyroidism and treated with Levothyroxine for at least 6 months
* Living independently in the community
* All TSH results within the range 0.4 - 4mU/L in the 3 months before commencing the study
* Participant has provided written informed consent for participation in the study, prior to any study-specific procedures

Exclusion Criteria:

* Established dementia and therefore deemed incapable of providing informed consent.
* Other medical conditions which, inthe opinion of the Chief Investigator, would prevent them from participating in the study (for example, end stage cancer, severe chronic health conditions where the patient is housebound)
* Nursing Homes or Residential Care Home residents
* Individuals with thyroid cancer: since they require high doses of LT4 to suppress their serum TSH
* Individuals on 25 mcg dailty of LT4: dose reduction will mean that they stop thyroid replacement treatment
* Non english speaking individuals
* Participation in any other investigational trials within the last 3 months
* Participants prescribed medications that can affect thyroid function (amiodarone, lithium, carbimazole or propylthiouracil)
* Known or suspected lactose intolerance (this would have implications for the proposed over-encapsulated IMP)

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Participant's acceptability of study design and willingness to enter study | Until completion of recruitment, approximately 24 months
  Participant's acceptability of study design as measured byt he completion rate of participants in each randomised group, as well as their willingness to enter the trial (consented participant to eligible participant approached ratio)

SECONDARY OUTCOMES:
Participant recruitment rate | Until completion of recruitment, approximately 24 months
  As measured by the number of patients randomised divided by the length of the recruitment period. The recruitment period runs from the date that recruitment opened to the date of last randomisation.
Time to achieve desired TSH levels | Until participant completion of SORTED 1 study, approximately within 24 weeks
  To review and assess the dose titration strategy (ie reduced LT4 dose or same dose LT4) and length of time required to achieved desired TSH levels (ie number of participants in each group that reach target TSH range at both 12 and 24 weeks)
Medication compliance | For the duration of participant involvment in the study, maximum of 25 weeks
  Tablet count
The acceptability of three patient completed questionnaires | For the duration of participant involvement in the study, maximum of 25 weeks
  The questionnaires include the generic QoL questionnaire (EQ-5D), validated disease-specific QoL questionanaire (ThyDQol) and disease specific hypothyroid-symptom check list (ThySC). The time taken to complete the three questionnaires will be recorded and questionnaire completion rates will be recorded and usefulnesss of questionnaires determined. Any third-party held required in a questionnaire's completion will be recorded.
Assessment of mobility | For the duration of participant involvement in this study, maximum of 25 weeks
  Measured by the nurse administered TUG Test, and the FRAT (Falls Risk Assessment Tool)
Change in specific cardiovascular risk factors | For the duration of participant involvement in the study, maximum of 25 weeks
  Lipid profile (total cholesterol, HDL, Triglycerides), blood pressure and body weight, and serum results
Measure of risk of falls | For the duration of participant involvement in the study, maximum 25 weeks
  Measure by nurse administrated FRAT (Falls Risk Assessment Tool) test.

CONTACTS AND LOCATIONS:
Overall Officials: Salman Razvi, Principal Investigator — Gateshead Health NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Bensham Hospital, Gateshead, Tyne and Wear
  - Clinical Research Facility, Newcastle upon Tyne, Tyne and Wear

REFERENCES:
- [Derived] Razvi S, Ingoe L, Ryan V, Pearce SH, Wilkes S. Study of Optimal Replacement of Thyroxine in the Elderly (SORTED) - results from the feasibility randomised controlled trial. Thyroid Res. 2016 Oct 10;9:5. doi: 10.1186/s13044-016-0034-x. eCollection 2016. PMID 27766119